CLINICAL TRIAL: NCT00586729
Title: Pilot Study to Evaluate Effectiveness of Vashe™ Wound Therapy as an Antimicrobial Irrigant in Burn Wound Management
Brief Title: Vashe Wound Therapy Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Valleywise Health (Other)
Collaborators: PuriCore, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007-012; 1200-0007
Record Dates: First submitted 2007-12-21; First posted 2008-01-04 (Estimated); Results first posted 2012-09-10 (Estimated); Last update posted 2012-09-14 (Estimated); Status verified 2012-09

CONDITIONS: Burns
Keywords: Burn; Burn wound management; Burn graft
MeSH Terms: conditions — Burns | interventions — Mafenide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vashe (Experimental): Vashe Wound Therapy applied to gauze dressing every 6 hours or as necessary to keep dressing moist for a total treatment duration of 5 days.
  Interventions: Device: Vashe
- 5% Mafenide Acetate (Active Comparator): 5% Mafenide Acetate applied to gauze dressing every 6 hours or as necessary to keep dressing moist for a total treatment duration of 5 days.
  Interventions: Drug: Mafenide acetate

INTERVENTIONS:
Device: Vashe — Antimicrobial irrigant
  Arms: Vashe
Drug: Mafenide acetate — Antimicrobial solution
  Arms: 5% Mafenide Acetate

SUMMARY:
This study will evaluate the efficacy, safety, and tolerability of topical Vashe™ Wound Therapy applied to gauze dressing every 6 hours or as necessary to keep dressing moist versus 5% Mafenide Acetate applied to gauze dressing every 6 hours or as necessary to keep dressing moist for a total treatment duration of 5 days.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 years and over requiring hospitalization for burn injury
* Burn injury requiring wound excision and auto-grafting
* Less than or equal to 20% Total Body Surface Area burns

Exclusion Criteria:

* Pregnant or lactating females
* Individuals with chlorine sensitivity
* Electrical, chemical and cold injury
* Burns to the face, hands, feet and or perineum area
* Steroid therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2009-07; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Foster, MD, Principal Investigator — District Medical Group
Locations (1):
- Maricopa Integrated Health System, Phoenix, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vashe | 5% Mafenide Acetate
Started | 14 | 9
Completed | 11 | 8
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vashe | 5% Mafenide Acetate | Total
Number analyzed (Participants) | 14 | 9 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 10 | 7 | 17
  >=65 years | 3 | 2 | 5
Age Continuous [Mean (Standard Deviation); unit: years] | 47.0 (17.9) | 52.7 (16.1) | 47.6 (17.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 10 | 6 | 16
Region of Enrollment [Number; unit: participants]
  United States | 14 | 9 | 23

OUTCOME MEASURES:

1. Secondary Outcome: Length of Stay
Description: Average hospital length of stay in days
Time Frame: 0 days, 3 days, 5 days and 14 days post-operation
Population: Per protocol
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Vashe | 5% Mafenide Acetate
Number analyzed (Participants) | 11 | 8
Days | 21.5 (4.2) | 15.6 (5.1)

2. Secondary Outcome: Hospital Cost Per Patient
Description: Average hospital irrigant cost per patient
Time Frame: Volume used from admission to discharge
Population: Per protocol
Measure: Mean (Standard Deviation); unit: Dollars
Arm/Group | Vashe | 5% Mafenide Acetate
Number analyzed (Participants) | 11 | 8
Dollars | 249.38 (93.43) | 393.00 (176.94)

3. Primary Outcome: Percentage of Grafted Area That is Viable at Day 14
Description: Percentage area of graft viability at 14 days as determined by clinical assessment of revascularization, adherence of the graft to the wound bed and color
Time Frame: 14 days
Population: Per protocol
Measure: Mean (Standard Deviation); unit: Percentage area
Arm/Group | Vashe | 5% Mafenide Acetate
Number analyzed (Participants) | 9 | 7
Percentage area | 96.3 (7.05) | 96.0 (3.83)

ADVERSE EVENTS:
Arm/Group | Vashe | 5% Mafenide Acetate
Serious Adverse Events (participants affected / at risk) | 2/11 | 1/8
Other Adverse Events (participants affected / at risk) | 11/11 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vashe (N=11) | 5% Mafenide Acetate (N=8)
MRSA infection (Infections and infestations) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vashe (N=11) | 5% Mafenide Acetate (N=8)
Hematological abnormality (Blood and lymphatic system disorders) | 6 | 5
Chemistry abnormality (Blood and lymphatic system disorders) | 7 | 7
Urinalysis abnormality (Renal and urinary disorders) | 10 | 7
UTI (Renal and urinary disorders) | 1 | 0
Vaginitis (Reproductive system and breast disorders) | 1 | 0
Possible seizure (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Change in affect (Psychiatric disorders) | 2 | 1
Coagulation abnormalities (Blood and lymphatic system disorders) | 2 | 1
Acute pain (Injury, poisoning and procedural complications) | 1 | 0
Chronic pain (Injury, poisoning and procedural complications) | 0 | 1
MRSA infection (Infections and infestations) | 1 | 0
Staph infection (Infections and infestations) | 1 | 0 — Not at test site
Cellulitis (Skin and subcutaneous tissue disorders) | 0 | 1
Surgical site drainage (Infections and infestations) | 0 | 1 — Not in test area
Vomiting (Gastrointestinal disorders) | 1 | 0
Fever (Metabolism and nutrition disorders) | 1 | 0
Chest pain (Cardiac disorders) | 0 | 1
Edema (Blood and lymphatic system disorders) | 0 | 1 — Not at test site
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Desaturation (Injury, poisoning and procedural complications) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Hypertrophic granulation tissue (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No